CLINICAL TRIAL: NCT02345889
Title: A 4-arm Randomized Controlled Trial of Fuse®, EndoCuff™, EndoRings™ and Standard Colonoscopy
Brief Title: A 4-arm Clinical Trial of Fuse®, EndoCuff™, EndoRings™ and Standard Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1412036333
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- FUSE® Colonoscopy (Active Comparator): A FUSE® system with 3 HD (high-definition) monitors will be used to perform the colonoscopy
  Interventions: Device: FUSE® Colonoscopy
- Colonoscopy with EndoCuff™ (Active Comparator): An EndoCuff™ distal attachment will be placed at the distal end of a standard colonoscope
  Interventions: Device: Colonoscopy with EndoCuff™
- Colonoscopy with EndoRings™ (Active Comparator): An EndoRings™ distal attachment will be placed at the distal end of a standard colonoscope
  Interventions: Device: Colonoscopy with EndoRings™
- Standard Colonoscopy (Active Comparator): A standard colonoscope will be used to complete the procedure
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: Colonoscopy with EndoCuff™ — colonoscopy performed with an EndoCuff™ device at the tip of a standard colonoscope
  Arms: Colonoscopy with EndoCuff™
Device: FUSE® Colonoscopy — colonoscopy performed with the FUSE® (full spectrum endoscopy) system
  Arms: FUSE® Colonoscopy
Device: Colonoscopy with EndoRings™ — colonoscopy performed with an EndoRings™ device at the tip of a standard colonoscope
  Arms: Colonoscopy with EndoRings™
Device: Standard Colonoscopy — Current standard of care colonoscopy
  Arms: Standard Colonoscopy

SUMMARY:
Adenoma detection rate (ADR) is a validated marker for reducing the risk of interval colorectal cancer after a screening colonoscopy. Recent studies suggest that novel devices attached to the colonoscope tip may improve the ADR of doctors performing a screening procedure

DETAILED DESCRIPTION:
Recent studies indicate that continuing medical education, time of colonoscopy during the day, forced longer withdrawal time, use of high definition colonoscopes all result in improving ADR although the gains have only been modest. To this end, adding novel devices to the tip of colonoscope may improve the ability of doctors to perform a better procedure. We therefore propose to identify the increase in ADR with 3 of these devices compared to standard colonoscopy. Fuse colonoscopy (2 cameras embedded at the side of the colonoscope tip providing an increased angle of view), EndoCuff (a plastic cap to fit the tip with flexible arms which hold the mucosa back aiding in inspection), EndoRings (similar to EndoCuff but the arms are wider) have been shown in tandem colonoscopy studies to improve the adenoma miss rates to 7-15% instead of the miss rates seen with standard colonoscopy which is usually about 40%. All these devices are FDA approved and are distributed in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Screening or Surveillance Colonoscopy

Exclusion Criteria:

* Personal history of Colorectal cancer or Inflammatory bowel disease
* Surgical resection of the colon or known colonic stricture
* Personal or family history of Polyposis syndromes or Lynch syndrome
* Referral for incomplete colonoscopy or known therapeutic polyp clearance
* Severe diverticular disease
* Referral for a positive hemoccult test in the past 6 months
* Known coagulopathy
* Inability to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1262 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Rex DK, Repici A, Gross SA, Hassan C, Ponugoti PL, Garcia JR, Broadley HM, Thygesen JC, Sullivan AW, Tippins WW, Main SA, Eckert GJ, Vemulapalli KC. High-definition colonoscopy versus Endocuff versus EndoRings versus full-spectrum endoscopy for adenoma detection at colonoscopy: a multicenter randomized trial. Gastrointest Endosc. 2018 Aug;88(2):335-344.e2. doi: 10.1016/j.gie.2018.02.043. Epub 2018 Mar 9. PMID 29530353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Started | 316 | 316 | 315 | 315
Completed | 295 | 299 | 295 | 299
Not Completed | 21 | 17 | 20 | 16
Not completed — Inadequate Bowel Prep | 17 | 16 | 18 | 14
Not completed — Polyposis identified during procedure | 1 | 1 | 0 | 1
Not completed — Recognized ineligible post-randomization | 1 | 0 | 2 | 1
Not completed — Ulcerative Colitis identified | 1 | 0 | 0 | 0
Not completed — Cecum not intubated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy | Total
Number analyzed (Participants) | 295 | 299 | 295 | 299 | 1188
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.3) | 63.2 (8.2) | 62.3 (7.9) | 62.3 (8.7) | 62.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 141 | 156 | 146 | 582
  Male | 156 | 158 | 139 | 153 | 606
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 272 | 276 | 276 | 269 | 1093
  Black or African American | 13 | 15 | 13 | 20 | 61
  Hispanic or Latino | 5 | 6 | 5 | 4 | 20
  Asian | 4 | 2 | 1 | 5 | 12
  Other | 1 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 1 | 1
Indication [Count of Participants; unit: Participants]
  Screening | 127 | 126 | 123 | 128 | 504
  Surveillance | 151 | 150 | 152 | 154 | 607
  Diagnostic | 16 | 23 | 20 | 16 | 75
  Unknown | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Adenomas Per Colonoscopy
Time Frame: During Procedure
Population: The number of adenomas was calculated overall for all three sites and then broken down into individual sites. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Mean (Standard Deviation); unit: Adenomas per Colonoscopy
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Adenomas per Colonoscopy
  All Sites | 1.53 (2.33) | 1.82 (2.58) | 1.55 (2.42) | 1.30 (1.96)
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 1.89 (2.69) | 2.17 (2.88) | 1.97 (2.77) | 1.59 (2.18)
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 0.83 (1.18) | 0.80 (1.25) | 0.72 (1.17) | 0.68 (1.19)
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 0.92 (1.15) | 2.00 (2.34) | 0.75 (0.94) | 0.80 (1.32)

2. Secondary Outcome: Number of Participants With Detected Adenoma
Time Frame: During Procedure
Population: The number of participants with detected adenomas was calculated overall for all three sites and then broken down into individual sites. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Participants
  All Sites | 166 | 191 | 167 | 154
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 117 | 137 | 127 | 115
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 37 | 35 | 29 | 28
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 12 | 19 | 11 | 11

3. Secondary Outcome: Percentage of Participants With Detected Adenoma
Time Frame: During Procedure
Population: The number of participants analyzed differed because the calculation was done for all three sites overall and then broken down into each specific site. Thus, only patients randomized to the treatment arm at that site were included in the specific site calculations instead of including the total number of patients randomized to that treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Percentage of Participants
  All Sites | 56 | 64 | 57 | 52
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 61 | 70 | 65 | 58
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 47 | 47 | 39 | 37
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 48 | 68 | 46 | 44

4. Secondary Outcome: Sessile Serrated Polyps Per Colonoscopy
Time Frame: During Procedure
Population: The number of sessile serrated polyps per colonoscopy was calculated overall for all three sites and then broken down into individual sites. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Mean (Standard Deviation); unit: Sessile Serrated Polyps per colonoscopy
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Sessile Serrated Polyps per colonoscopy
  All Sites | 0.17 (0.54) | 0.17 (0.54) | 0.20 (0.81) | 0.18 (0.74)
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 0.24 (0.64) | 0.23 (0.63) | 0.29 (0.98) | 0.25 (0.89)
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 0.03 (0.16) | 0.04 (0.26) | 0.01 (0.12) | 0.03 (0.16)
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 0.04 (0.20) | 0.07 (0.26) | 0.04 (0.20) | 0.04 (0.20)

5. Secondary Outcome: Number of Participants With Detected Sessile Serrated Polyp
Description: Number of patients with 1 or more sessile serrated polyps
Time Frame: During Procedure
Population: The number of participants with detected sessile serrated polyps was calculated overall for all three sites and then broken down into individual sites. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Participants
  All Sites | 36 | 33 | 33 | 30
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 33 | 29 | 31 | 27
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 2 | 2 | 1 | 2
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 1 | 2 | 1 | 1

6. Secondary Outcome: Percentage of Participants With Detected Sessile Serrated Polyp
Time Frame: During Procedure
Population: The number of participants analyzed for each site differed because the percentage of patients with a sessile serrated polyp was calculated specifically for the site. Thus, only patients randomized to the treatment arm at that site were included in the calculation instead of including the total number of patients randomized to the treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Percentage of Participants
  All Sites | 12 | 11 | 11 | 10
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 17 | 15 | 16 | 14
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 3 | 3 | 1 | 3
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 4 | 7 | 4 | 4

7. Secondary Outcome: Number of Participants With a Detected Polyp
Time Frame: During Procedure
Population: The number of participants with a detected polyp was calculated overall for all three sites and then broken down into individual sites. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Participants
  All Sites | 226 | 247 | 231 | 212
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 162 | 175 | 171 | 155
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 46 | 50 | 42 | 38
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 18 | 22 | 18 | 19

8. Secondary Outcome: Percentage of Participants With a Detected Polyp
Time Frame: During Procedure
Population: The number of participants analyzed for each site differed because the percentage of patients with a polyp was calculated for each site specifically. Thus, only patients randomized to the treatment arm at that site were included in the calculation instead of including the total number of patients randomized to the treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Percentage of Participants
  All Sites | 77 | 83 | 78 | 71
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 84 | 89 | 87 | 78
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 59 | 68 | 56 | 51
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 72 | 79 | 75 | 76

9. Secondary Outcome: Cecal Insertion Time
Time Frame: During Procedure
Population: The mean insertion time was calculated overall for all three sites and then broken down into individual sites. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Seconds
  All Sites | 422 (319) | 354 (216) | 403 (263) | 468 (311)
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 366 (243) | 320 (179) | 352 (191) | 395 (225)
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 642 (405) | 503 (254) | 581 (356) | 731 (385)
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 170 (62) | 193 (93) | 251 (110) | 242 (80)

10. Secondary Outcome: Cecal Insertion Times When no Gastroenterology Fellow Was Involved in Insertion
Time Frame: During Procedure
Population: Gastroenterology fellows were allowed to assist in inserting the scope, but times included in this analysis were from insertions done completely by the physician. This is why the overall number analyzed differs from the number analyzed in other outcome measure as well as why the numbers differ depending on site and randomization arm.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 173 | 169 | 173 | 176
Seconds
  All Sites | 320 (256) | 265 (173) | 331 (222) | 380 (252)
  Indianapolis: number analyzed (Participants) | 114 | 114 | 119 | 127
  Indianapolis | 283 (185) | 239 (127) | 277 (127) | 340 (169)
  Milan: number analyzed (Participants) | 34 | 28 | 32 | 25
  Milan | 556 (378) | 438 (269) | 588 (345) | 718 (401)
  New York: number analyzed (Participants) | 25 | 27 | 22 | 24
  New York | 170 (62) | 193 (93) | 251 (110) | 242 (80)

11. Secondary Outcome: Inspection Time
Time Frame: During Procedure
Population: The mean inspection time of all three sites overall was calculated as well as the mean inspection time for each individual site. The number of participants in each arm differed at each site, which is why the number analyzed differs depending on site and randomization.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Seconds
  All Sites | 444 (103) | 419 (95) | 417 (147) | 421 (112)
  Indianapolis: number analyzed (Participants) | 192 | 197 | 196 | 199
  Indianapolis | 418 (91) | 392 (89) | 388 (160) | 378 (83)
  Milan: number analyzed (Participants) | 78 | 74 | 75 | 75
  Milan | 501 (109) | 492 (78) | 484 (92) | 522 (120)
  New York: number analyzed (Participants) | 25 | 28 | 24 | 25
  New York | 467 (95) | 414 (84) | 438 (96) | 454 (81)

12. Secondary Outcome: Number of Conventional Adenomas by Size in the Right Side of the Colon, Which Includes the Cecum, Ascending Colon, and Hepatic Flexure.
Time Frame: During Procedure
Measure: Number; unit: Adenomas
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Adenomas
  All | 205 | 253 | 213 | 194
  1-5mm | 160 | 199 | 162 | 145
  6-9mm | 28 | 37 | 31 | 35
  greater than or equal to 10mm | 17 | 17 | 20 | 14

13. Secondary Outcome: Percent of Conventional Adenomas by Size in the Right Side of the Colon, Which Includes the Cecum, Ascending Colon, and Hepatic Flexure.
Time Frame: During Procedure
Measure: Number; unit: Percentage of Adenomas
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Percentage of Adenomas
  1-5mm | 78 | 79 | 76 | 75
  6-9mm | 14 | 15 | 15 | 18
  greater than or equal to 10mm | 7 | 7 | 9 | 7

14. Secondary Outcome: Number of Sessile Serrated Polyps by Size in the Right Side of the Colon, Which Includes the Cecum, Ascending Colon, and Hepatic Flexure.
Time Frame: During Procedure
Measure: Number; unit: Sessile Serrated Polyps
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Sessile Serrated Polyps
  All | 20 | 32 | 29 | 25
  1-5mm | 9 | 11 | 8 | 9
  6-9mm | 6 | 10 | 8 | 4
  greater than or equal to 10mm | 5 | 11 | 13 | 12

15. Secondary Outcome: Percent of Sessile Serrated Polyps in the Right Side of the Colon, Which Includes the Cecum, Ascending Colon, and Hepatic Flexure.
Time Frame: During Procedure
Measure: Number; unit: Percentage of Sessile Serrated Polyps
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
Number analyzed (Participants) | 295 | 299 | 295 | 299
Percentage of Sessile Serrated Polyps
  1-5mm | 45 | 34 | 28 | 36
  6-9mm | 30 | 31 | 28 | 16
  greater than or equal to 10mm | 25 | 34 | 45 | 48

ADVERSE EVENTS:
Time Frame: 28 months
Arm/Group | Standard Colonoscopy | Colonoscopy With EndoCuff™ | Colonoscopy With EndoRings™ | FUSE® Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/295 | 0/299 | 0/295 | 0/299
Serious Adverse Events (participants affected / at risk) | 0/295 | 0/299 | 0/295 | 0/299
Other Adverse Events (participants affected / at risk) | 0/295 | 0/299 | 0/295 | 0/299

LIMITATIONS AND CAVEATS:
* Recruitment was uneven across the sites, and there were some differences between sites with regard to detection. Thus, some caution is appropriate in concluding generalizability.
* Endoscopists were not blinded to which device was in use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT02345889/Prot_SAP_000.pdf